CLINICAL TRIAL: NCT04972292
Title: A Clinical, Multicenter, Randomized, Parallel-group, Double-blind, Double-dummy, Comparative Study of Non-inferiority of the Fixed Dose Combination of Codeine 30 Mg/dipyrone 500 Mg from Eurofarma Versus Tylex® (codeine 30 Mg/paracetamol 500 Mg) in the Treatment of Moderate to Intense Pain Post-impacted Third Lower Molar Extraction
Brief Title: Fixed Dose Combination of COdeine + DIpyrone to Mitigate Moderate to Intense Pain Post-impacted Third Lower Molar Extraction
Acronym: CODI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF174
Record Dates: First submitted 2021-07-15; First posted 2021-07-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pain
Keywords: postoperative; third lower molar extraction
MeSH Terms: conditions — Pain | interventions — Dipyrone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: FDC of codeine 30 mg/dipyrone 500 mg from Eurofarma Laboratórios SA (Experimental): Subjects randomized to this group will receive one (1) experimental drug tablet + one (1) Tylex® placebo tablet when the postoperative pain becomes moderate to intense (≥ 40 mm at a VAS of 0-100 mm). Then, subjects will be instructed to use the study treatment whenever it is necessary for pain relief, respecting a minimal interval of six (6) hours between two administrations, for up to 3 days (72 hours after the initial dose).
  Interventions: Drug: FDC of codeine 30 mg/dipyrone 500 mg
- Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg) (Active Comparator): Subjects randomized to this group will receive one (1) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (1) FDC placebo tablet when the postoperative pain becomes moderate to intense (≥ 40 mm at a VAS of 0-100 mm). Then, subjects will be instructed to use the study treatment whenever it is necessary for pain relief, respecting a minimal interval of six (6) hours between two administrations, for up to 3 days (72 hours after the initial dose).
  Interventions: Drug: Tylex

INTERVENTIONS:
Drug: FDC of codeine 30 mg/dipyrone 500 mg — Group 1: receive one (1) experimental drug tablet (FCD of codeine 30mg/dipyrone 500mg) + one (1) Tylex® placebo.
  Arms: Group 1: FDC of codeine 30 mg/dipyrone 500 mg from Eurofarma Laboratórios SA
Drug: Tylex — Group 2: receive one (1) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (1) FDC placebo tablet
  Arms: Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg)

SUMMARY:
A clinical, multicenter, randomized, parallel-group, double-blind, double-dummy, comparative study of non-inferiority.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
Subjects aged between 16 and 35 years old, with indicated surgical removal of impacted third lower molar, will be randomized at a 1:1 ratio to receive the FDC of codeine 30 mg/dipyrone 500 mg from Eurofarma Laboratórios SA (experimental drug) or the FDC of codeine 30 mg/paracetamol 500 mg (Tylex® - Janssen-Cilag Farmacêutica Ltda) as tablets for up to three (3) days. Subjects whose surgery lasts no more than 40 minutes and showing moderate to intense postoperative pain up to four (4) hours after surgery will be randomized. The first study drug administration will take place at the clinical investigation site when the postsurgical pain becomes moderate/intense (≥ 40 mm at a visual analogue scale [VAS] of 0-100 mm). Then, subjects will be instructed to use the study treatment whenever it is necessary for pain relief, respecting a minimal interval of six (6) hours between two administrations, for up to three (3) days (72 hours after the initial dose). Subjects will evaluate the pain relief using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) in 1-hour intervals (1, 2, 3, 4, 5 and 6h). The sum of the relief scores over 6 hours determines the TOTPAR6

Subjects who meet all of the eligibility criteria will be randomized to one of the following treatment groups:

Group 1: FDC of codeine 30 mg/dipyrone 500 mg from Eurofarma Laboratórios SA (experimental drug) - Subjects randomized to this group will receive one (1) experimental drug tablet + one (1) Tylex® placebo tablet when the postoperative pain becomes moderate to intense (≥ 40 mm at a VAS of 0-100 mm).

Group 2: Tylex® (codeine 30 mg/paracetamol 500 mg) - Subjects randomized to this group will receive one (1) Tylex® tablet (codeine 30 mg/paracetamol 500 mg) + one (1) FDC placebo tablet when the postoperative pain becomes moderate to intense (≥ 40 mm at a VAS of 0-100 mm).

The subjects will be allowed to use the rescue medication if necessary: Paracetamol 500 mg (Tylenol® 500 mg).

All subjects must have three (3) on-site visits at the research site. Three (3) phone calls will take place between the on-site visits: Screening visit (Vs), randomization visit (Vr), first phone call (CT1), second phone call (CT2), third phone call (CT3), final visit (Vf).

The period for including subjects in the study will start after the required ethical and regulatory approvals and its estimated duration will be of up to 12 months. The approximate study duration will be of 9 ± 2 days for each subject.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 16 and 35 years old (inclusive).
2. Presence of impacted third lower molar with surgical removal indicated (diagnosed via panoramic x-ray within six [6] months before inclusion in the study), at vertical, mesioangular or horizontal position as per the Winter's classification, provided that it belongs to the following Pell & Gregory's classes:
3. Maximum surgery duration of 30 minutes, counted from the initial incision to the impacted third molar extraction.
4. Moderate to intense postoperative pain (≥ 40 mm at a VAS of 0-100 mm) up to four (4) hours after the end of the surgery (counted from the end of the suture).
5. Informed Consent Form (ICF) and Informed Assent Form (IAF) signature, when applicable, before performing any study procedure.

Exclusion Criteria:

1. Known hypersensitivity to dipyrone or to other pirazolones or pirazolidines (e.g.: phenazone, propyphenazone, isopropylaminophenazone, phenylbutazone, oxyphenbutazone), including history of previous agranulocytosis with one of these substances;
2. Known hypersensitivity to codeine or to other opioid agents;
3. Known hypersensitivity to paracetamol or to any component of the Tylex® formulation;
4. Bone marrow function impairment (e.g.: after cytostatic treatment) or hematopoietic system diseases;
5. History of bronchospasm or other anaphylactoid reactions (e.g.: hives, rhinitis, angioedema) associated with the use of analgesics, such as salicylates, paracetamol, diclofenac, ibuprofen, indomethacin, naproxen;
6. History of significant hypotensive reaction associated with the administration of dipyrone;
7. Abuse of illegal drugs, including alcoholism; emotional instability and/or previous attempt of suicide;
8. Pregnancy or breastfeeding.
9. Women of childbearing potential who do not agree to use a known effective birth control method, unless the participants are surgically sterile or state they are expressly free of the risk of getting pregnant for not having sexual intercourse or for having sexual intercourse with no reproductive potential.
10. Participation in a clinical research protocol within the past 12 months, unless the investigator considers that the participation in the study could result in a direct benefit to the subject.
11. Presence of any condition that, in the investigator's opinion, would make the subject ineligible to participate in the study.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
sum of pain relief scores over 6 hours (TOTPAR6) | 6 hours
  After the first study treatment dose is given, subjects will evaluate the pain relief using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) in 1-hour intervals (1, 2, 3, 4, 5 and 6 hours). The sum of the relief scores over 6 hours determines the TOTPAR6, which ranges from 0 to 24, with a higher score indicating more pain relief.

SECONDARY OUTCOMES:
Sum of pain relief scores over four (4) hours (TOTPAR4) | 4 hours
  After the first study treatment dose is given, subjects will evaluate the pain relief using a 5-point categorical scale (0 = no relief, 1 = little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief) in 1-hour intervals (1, 2, 3, 4 hours)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Eurofarma Laboratórios S.A, Brasil, São Paulo
  - Eurofarma Laboratorios S.A, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No